CLINICAL TRIAL: NCT03972943
Title: Modulation of Morbidity and Disease Progression in Polycythemia Vera (PV) and Essential Thrombocythemia (ET) Patients With Obstructive Sleep Apnea (OSA) by CPAP
Brief Title: CPAP in Treating Obstructive Sleep Apnea in Patients With Polycythemia Vera or Essential Thrombocythemia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study terminated due to lack of funding
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI114917; NCI-2019-01690 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCI114917 (Other: Huntsman Cancer Institute/University of Utah); P30CA042014 (NIH)
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: CALR Gene Mutation; Essential Thrombocythemia; JAK2 Gene Mutation; MPL Gene Mutation; Obstructive Sleep Apnea Syndrome; Polycythemia Vera
MeSH Terms: conditions — Thrombocythemia, Essential; Sleep Apnea, Obstructive; Polycythemia Vera | interventions — Continuous Positive Airway Pressure; Watchful Waiting; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (observation) (Active Comparator): Patients not diagnosed with OSA undergo observation for 6 months.
  Interventions: Other: Patient Observation; Other: Questionnaire Administration
- Cohort II: (CPAP treatment) (Experimental): Patients diagnosed with OSA and prescribed a CPAP machine for treatment receive continuous treatment with CPAP for 6 months.
  Interventions: Procedure: Continuous Positive Airway Pressure; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Continuous Positive Airway Pressure — Receive CPAP treatment
  Other Names: Continuous positive airway pressure (CPAP); CPAP
  Arms: Cohort II: (CPAP treatment)
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; observation; Watchful Waiting
  Arms: Cohort I (observation)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I trial studies how well the use of a continuous positive airway pressure (CPAP) machine works in treating obstructive sleep apnea in patients with polycythemia vera or essential thrombocythemia. Obstructive sleep apnea is a condition where a person stops breathing during sleep, and is estimated to affect 30 to 50 percent of patients with polycythemia vera or essential thrombocythemia. A patient with obstructive sleep apnea typically snores, has disrupted sleep, experiences morning headaches, and has daytime sleepiness. Patients diagnosed with obstructive sleep apnea are typically treated with a device called CPAP. The CPAP provides pressurized air that keeps upper air passages open during sleep and may prevent them from narrowing or collapsing as occurs during snoring or sleep apnea.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To understand effects of continuous positive airway pressure (CPAP) for obstructive sleep apnea (OSA) on the course of polycythemia vera/essential thrombocythemia (PV/ET).

EXPLORATORY OBJECTIVES:

I. To estimate prevalence of OSA in patients with myeloproliferative neoplasms. II. To understand effects of CPAP for sleep apnea on the course of myeloproliferative neoplasms (MPNs).

III. To correlate OSA severity with thrombotic and inflammatory marker values in patients with PV/ET at baseline.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I (OBSERVATIONAL COHORT): Patients not diagnosed with OSA undergo observation for 6 months.

COHORT II (TREATMENT COHORT): Patients diagnosed with OSA and prescribed a CPAP machine for treatment receive continuous treatment with CPAP for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* OSA SCREENING ELIGIBILITY CRITERIA: Documented diagnosis of essential thrombocythemia or polycythemia vera by either 2008 WHO criteria or 2016 WHO Criteria prior to screening.
* OSA SCREENING ELIGIBILITY CRITERIA: For subjects receiving therapy for PV or ET (i.e. hydroxyurea, peginterferon, etc.): Patients must be on a stable dose for >= 28 days prior to study entry and expected to remain on a stable dose for the duration of trial participation. It is anticipated that during the 6 month duration of study, there will not be any dose modification of hydroxyurea or interferon and this will be communicated to treating providers and patient during enrollment into the trial. However, clinically indicated dose modification of PV/ET therapy while on trial will not necessitate CPAP study discontinuation.
* OSA SCREENING ELIGIBILITY CRITERIA: Subject must have =< 20.0 pack-year smoking history OR have quit smoking => 3 years ago and do not have any current symptoms of COPD and/or have normal pulmonary function tests.
* OSA SCREENING ELIGIBILITY CRITERIA: Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* OSA SCREENING ELIGIBILITY CRITERIA: Negative serum or urine pregnancy test at screening for women of childbearing potential.
* OSA SCREENING ELIGIBILITY CRITERIA: Highly effective contraception for both male and female subjects from study enrollment through treatment, and for at least 3 months after last study treatment administration if the risk of conception exists.
* OSA SCREENING ELIGIBILITY CRITERIA: Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* OSA SCREENING ELIGIBILITY CRITERIA: Able to read and complete required study questionnaires.
* TREATMENT ELIGIBILITY CRITERIA: Eligible for OSA Screening Component portion of this trial.
* TREATMENT ELIGIBILITY CRITERIA: Diagnosed OSA with Sleep Study score >= 5.
* TREATMENT ELIGIBILITY CRITERIA: Snoring, Tiredness, Observed Apnea, Blood Pressure, Body Mass Index, Age, Neck Circumference and Gender (STOP-BANG) screening questionnaire score >= 3.
* TREATMENT ELIGIBILITY CRITERIA: Willingness to comply with required CPAP compliance rate of >= 4hrs/day for 70% of days over 6 months of CPAP treatment.
* TREATMENT ELIGIBILITY CRITERIA: Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* OSA SCREENING ELIGIBILITY CRITERIA: Use of JAK2 inhibitors within 6 months prior to registration.
* OSA SCREENING ELIGIBILITY CRITERIA: Previous or current use of TNF inhibitors.
* OSA SCREENING ELIGIBILITY CRITERIA: Prior substantial, prolonged use of CPAP or alternative therapy for OSA, including oxygen. No more than 6 monthsof continuous therapy with CPAP in the last 5 years will be allowed.
* OSA SCREENING ELIGIBILITY CRITERIA: Autoimmune disease requiring concurrent use of immunomodulatory, including rheumatologic disorders.
* OSA SCREENING ELIGIBILITY CRITERIA: Prior invasive cancer (except nonmelanoma skin cancer) unless disease free for at least 2 years or life expectancy without treatment is greater than 2 years, e.g., low risk localized prostate cancer.
* OSA SCREENING ELIGIBILITY CRITERIA: The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months of screening. Patients receiving anti-coagulant therapy for previous thromboembolic event will be allowed to enroll on study.
  * Other clinically significant disorders that would preclude safe study participation.

    * End stage Renal disease
    * Advanced liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
    * Active (acute or chronic) or uncontrolled severe infection
* OSA SCREENING ELIGIBILITY CRITERIA: Known history of human immunodeficiency virus (HIV), chronic hepatitis B virus (HBV), or hepatitis C virus (HCV) infection.
* TREATMENT ELIGIBILITY CRITERIA: Use of JAK2 inhibitors within 6 months of registration.
* TREATMENT ELIGIBILITY CRITERIA: Previous or current use of TNF inhibitors.
* TREATMENT ELIGIBILITY CRITERIA: Prior use of CPAP or alternative therapy for OSA, including oxygen.
* TREATMENT ELIGIBILITY CRITERIA: Autoimmune disease requiring concurrent use of immunomodulatory, including rheumatologic disorders.
* TREATMENT ELIGIBILITY CRITERIA: Prior invasive cancer (except nonmelanoma skin cancer) unless disease free for at least 2 years or life expectancy without treatment is greater than 2 years, e.g., low risk localized prostate cancer.
* TREATMENT ELIGIBILITY CRITERIA: The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months of screening. Patients receiving anti-coagulant therapy for previous thromboembolic event will be allowed to enroll on study.
  * Other clinically significant disorders that would preclude safe study participation.

    * End stage Renal disease
    * Advanced liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
    * Active (acute or chronic) or uncontrolled severe infection
* TREATMENT ELIGIBILITY CRITERIA: Known history of HIV, chronic hepatitis B virus (HBV), or hepatitis C virus (HCV) infection.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Change in Myeloproliferative Neoplasm Symptom Assessment Form - Total Symptom Score (MPN-SAF TSS) | Baseline, after 3 months, and after 6 months on trial
  Will be tested at the two-sided 0.025 significance level to provide overall control of the type I error for the co-primary endpoints at 0.05. The endpoints will be summarized by mean, median, range, standard deviation, interquartile range and boxplots. Scatterplots will be used to show bivariate associations. An assessment of normality will be made prior to statistical testing. Paired t tests will be used to analyze endpoints that are sufficiently Gaussian in distribution. Paired Wilcoxon tests will be used to analyze variables that are highly skewed or otherwise non-Gaussian in distribution.
Change in JAK2 V617F allele burden | Baseline, after 3 months, and after 6 months on trial
  Will be tested at the two-sided 0.025 significance level to provide overall control of the type I error for the co-primary endpoints at 0.05. The endpoints will be summarized by mean, median, range, standard deviation, interquartile range and boxplots. Scatterplots will be used to show bivariate associations. An assessment of normality will be made prior to statistical testing. Paired t tests will be used to analyze endpoints that are sufficiently Gaussian in distribution. Paired Wilcoxon tests will be used to analyze variables that are highly skewed or otherwise non-Gaussian in distribution.

OTHER OUTCOMES:
Proportion of patients with a diagnosis of obstructive sleep apnea (OSA) | During the OSA screening
  Assessed by Snoring, Tiredness, Observed Apnea, Blood Pressure, Body Mass Index, Age, Neck Circumference and Gender (STOP-BANG) questionnaire. The proportion of patients whose results indicate a diagnosis of OSA will be calculated. All patients with a diagnosis of OSA, regardless of whether they are enrolled to the treatment component of the study, will be counted towards the assessment of prevalence. An assessment of normality will be made prior to statistical testing. Paired t tests will be used to analyze endpoints that are sufficiently Gaussian in distribution. Paired Wilcoxon tests will be used to analyze variables that are highly skewed or otherwise non-Gaussian in distribution.
Leucocytes, platelets, red cell counts, and tumor necrosis factor (TNF) analysis | Baseline, after 3 months, and after 6 months on trial
  The endpoints will be summarized by mean, median, range, standard deviation, interquartile range and boxplots. Scatterplots will be used to show bivariate associations. An assessment of normality will be made prior to statistical testing. Paired t tests will be used to analyze endpoints that are sufficiently Gaussian in distribution. Paired Wilcoxon tests will be used to analyze variables that are highly skewed or otherwise non-Gaussian in distribution.
Thrombotic and inflammatory marker levels for all patients | Baseline, after 3 months, and after 6 months on trial
  Will be measured in blood samples taken from all patients. OSA-related adverse events reported in the Treatment Cohort at these timepoints will be correlated with these marker levels. Pearson or Spearman correlation will be used to assess correlation between thrombo-inflammatory markers and oximetric abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Sundar, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (2):
- United States (2):
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Veterans Administration Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No